CLINICAL TRIAL: NCT00522119
Title: Genetic and Functional Analyses of Chromosome 1 Hypertension Susceptibility
Brief Title: Analysis of Genes That Predispose People to Develop High Blood Pressure
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Yen-Pei Christy Chang, PI, University of Maryland, Baltimore
Other Study IDs: 1403; R01HL088120 (NIH)
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Hypertension
Keywords: Essential Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — For each subject, blood and urine samples were collected at various time points during for interventions designed to study cardiovascular biology, including (1) a high-fat challenge, after which we measured the post-prandial excursion in triglycerides; (2) a cold pressor stress test (CPT), for which we measured changes in blood pressure and endothelial function; (3) a dietary salt intervention, involving 6-day ingestion of a high-salt diet, followed by 6-day ingestion of a low-salt diet, during which we measured changes in blood pressure; and (4) 14 days of low-dose aspirin therapy, during which we measured changes in platelet function. The exact protocol is published in the American Heart Journal, Volume 155, Issue 5, May 2008, pages 823-828.
Oversight: Data Monitoring Committee: No

SUMMARY:
High blood pressure affects nearly one third of all individuals in the United States. It is believed that genetic factors may predispose some people to develop this disease. This study will identify and characterize variations in three genes known to play a part in the development of high blood pressure.

DETAILED DESCRIPTION:
High blood pressure is one of the most common health problems in this country. It can be caused by many factors, including stress, diet, diabetes, kidney disease, or obesity. In many people, there is no identifiable cause for their high blood pressure. If high blood pressure goes untreated, it can lead to heart failure, kidney failure, or stroke. Previous studies have shown that variations in three genes in chromosome 1-ATP1B1, RGS5, and SELE-cause some people to be more susceptible to developing high blood pressure. All three of these genes are involved in the development of proteins that play a role in regulating blood pressure, but it is not known exactly how variations in these genes affect blood pressure levels. This study will examine previously collected genetic samples from participants in two studies, the GenNet study and the Heredity and Phenotype Interaction (HAPI) Heart study. Study researchers will analyze the samples to identify and characterize variations in the ATP1B1, RGS5, and SELE genes. Results from this study may lead to more effective diagnostic and treatment options for people with high blood pressure.

ELIGIBILITY:
Inclusion criteria:

* Amish individuals from the Lancaster community in PA.

Study-wide Exclusion criteria:

* Age< 20 yrs
* Non-Amish descent
* Currently pregnant or postpartum <6 m
* Blood pressure at the time of screening >180/105 (SBB/DBP) mm Hg
* Prescription medication use potentially affecting outcomes and vitamin or over-the-counter remedies that cannot be willingly or safely discontinued from 1 week before protocol initiation and until the end of the study (ie, β-blockers; calcium channel antagonists; ACE inhibitors; diuretics; lipid-lowering agents; nitrates; systemic glucocorticoids; adrenergic or cholinergic-acting agents, including cold formulas and antidepressants; and diet-weight loss agents)
* Coexisting malignancy
* Serum creatinine>2.0 mg/dL
* AST or ALT >twice the upper limit of normal
* Hematocrit <32%
* TSH <0.4 or >5.5 mIU/L

Intervention-specific exclusion criteria:

* Cold pressor stress test: history of Raynaud's disease
* High-fat challenge: malabsorption disorders, lactose intolerance, symptoms of gallbladder disease, and/or history of pancreatitis
* Dietary salt intervention: stage III or greater congestive heart failure and/or allergies to foods in the diet
* Aspirin intervention: history of bleeding disorder, gastrointestinal bleeding, blood pressure at the time of screening >160/95 mm Hg, current use of aspirin for a condition that would place the subject at increased risk if it were to be discontinued for 14 days before protocol initiation (eg, history of unstable angina, myocardial infarction, angioplasty, coronary artery bypass grafting, atrial fibrillation, stroke or transient ischemic attack, type 2 diabetes, or deep vein thrombosis/other thrombosis), polycythemia (hematocrit >52%), thrombocytosis (platelet count > 500 000), thrombocytopenia (platelet count <75 000), surgery within the last 6 months, aspirin allergy, current breastfeeding, and/or aggregation with collagen 5 μg/mL <6.65 Ω or >26 Ω or no aggregation at baseline with arachidonic acid

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Characteristic Men (n = 460) Women (n = 408) Age (y) 42.2 ± 0.6 45.4 ± 0.7 BMI (kg/m2) 25.6 ± 0.1 27.8 ± 0.3 TCHOL (mg/dL) 202.5 ± 2.1 215.7 ± 2.5 HDL (mg/dL) 52.6 ± 0.6 59.5 ± 0.8 TG (mg/dL) 63.9 ± 1.7 73.8 ± 2.3 SBP (mm Hg) 121.5 ± 0.6 121.4 ± 0.8 DBP (mm Hg) 77.6 ± 0.4 75.8 ± 0.4 Diabetes (%) 0.9 1.0 Current smokers (%) 20.0 0.0
  * on lipid-lowering medications 1.1 1.0
  * on antihypertensive medications 0.2 0.3
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2006-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yen Pei C. Chang, PhD, Principal Investigator — University of Maryland, Baltimore

REFERENCES:
- See also: Click here for the HAPI Heart Study Web site — https://www.medschool.umaryland.edu/endocrinology/Amish-Research-Program/Selected-Amish-Studies/Heredity--Phenotype-Interaction-Heart-Study-HAPI/